CLINICAL TRIAL: NCT02802332
Title: Use of a Foot Length Card to Improve Careseeking Practices of Vulnerable Newborns in Sarlahi District, Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Save the Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00085037
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Low Birth Weight Babies; Preterm Babies
Keywords: neonatal; preterm; Nepal; family-initiated identification; basic newborn care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Footlength Card (Active Comparator): Pregnant women will receive a card that enables them to measure the length of their baby's foot. The card contains a phone number to pre-recorded message that provides basic information/advice regarding care of preterm and/or low birth weight babies
  Interventions: Behavioral: Footlength Card
- No Footlength Card (No Intervention): Women in this group do receive any footlength card.

INTERVENTIONS:
Behavioral: Footlength Card — The footlength card has an image of a baby's foot. The card is to be held up against the baby's foot after birth; if a baby's foot is smaller than the image, or if the woman/family member is concerned about the health of their baby, they can call the number printed on the card and hear a pre-recorded message about basic care for newborn babies
  Arms: Footlength Card

SUMMARY:
This study will evaluate whether or not provision of a simple card ("footlength card") that allows identification of low birth weight and/or preterm babies through measurement of the length of a baby's foot, can improve basic newborn care behaviors in rural Nepal.

DETAILED DESCRIPTION:
This study will evaluate a recently developed, simple, low-cost tool that can help recently delivered women and their family members identify whether or not their newborn baby needs extra care/attention. Some prior studies of the relationship between anthropometric measures (such as chest-circumference, footlength, head circumference, etc) and preterm birth or low birth weight, have shown that these measures can be used to identify high-risk/vulnerable babies. One such measure, foot length, has been shown to be a reasonable tool, and one that can be simply performed by mothers, without disturbing the newborn infant. With this in mind, Save The Children has developed a low cost card with an image of a baby's foot on one side, along with a toll-free number and some key messages on how to use the card. Specifically, pregnant women can be given this card during an antenatal contact, along with some basic instructions on its use. Then, after their baby is born, the newly delivered woman, other family member, or low-level facility provider can compare the length of the baby's foot to the image on the card, by lining the baby's foot up with the card. If the baby's foot is shorter than the image on the card, a toll-free number (provided on the card itself) can be used to access a set of standardized messages about how to take care of the baby.

In this proposed study, Save the Children, Johns Hopkins University (JHU), and the JHU-led Nepal Nutrition Intervention Project - Sarlahi (NNIPS) will give this card to women currently enrolled in the Nepal Oil Massage Study (NCT01177111), explain its use, follow up with the woman after delivery to determine if she used the card, and query her about her experience using the card, calling the toll-free number, and recalling the messages given. Additionally, one of the NNIPS staff workers will use the same card to measure the baby's foot. Ultimately, the study will summarize women's experience using this card, and provide guidance to Save the Children, the Ministry of Health and Population (MOHP), and other stakeholders regarding future programmatic scale up of the use of this card.

ELIGIBILITY:
Inclusion Criteria:

* Woman is pregnant
* Woman is enrolled in ongoing newborn oil massage study

Exclusion Criteria:

* Not pregnant
* Not enrolled in ongoing newborn oil massage study

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4574 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
skin to skin contact | within first 28 days after birth
  Does the mother report practicing skin to skin contact during the first 28 days after birth
careseeking for newborn | within first 28 days after birth
  Does the mother report seeking care for newborn (either routine postnatal care OR careseeking for illness) during the first 28 days after birth

CONTACTS AND LOCATIONS:
Overall Officials: Luke C Mullany, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Nepal Nutrition Intervention Project, Hariaun, Sarlahi District, Nepal

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data

REFERENCES:
- [Derived] Hodgins S, Rajbhandari B, Joshi D, Ban B, Khatry S, Mullany LC. Community-based cluster randomized controlled trial: empowering households to identify and provide appropriate care for low-birthweight newborns in Nepal. BMC Public Health. 2020 Aug 24;20(1):1274. doi: 10.1186/s12889-020-09317-w. PMID 32838783